CLINICAL TRIAL: NCT03243565
Title: Effect of Vaxoral® (OM-85) on Frequency of Respiratory Tract Infections and Size of Adenoid Tissue in Preschool Children With Adenoid Hypertrophy
Brief Title: Effect of OM-85 on Respiratory Tract Infections and Adenoid Tissue in Children With Adenoid Hypertrophy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Serap Ozmen, MD, Pediatric Allergist and Assoc. Prof of Pediatrics, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17-AKD-2
Record Dates: First submitted 2017-07-26; First posted 2017-08-09 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Adenoid Hypertrophy; Adenoid Hyperplasia; Respiratory Tract Infections; Preschool Children
Keywords: adenoid hypertrophy; Adenoid Hyperplasia; children; respiratory tract infection; adenotonsillectomy; OM-85
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: A randomised, double-blind, placebo-controlled, parallel group, phase IV study. First group will receive OM-85 (first 10 day consecutive 3 months; standard treatment regimen) Second group will receive matching placebo at the same posology (first 10 day consecutive 3 months).
  A second cure of treatment will be given 6 months after inclusion. Patients will be recruited from 01 August 2017 to 01 February 2018. The trial will begin in August 2017 and will be completed in February 2019.
  By this way every patient will be studied over all seasons (1 year study) .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by throwing the coin. Family of patients and doctor (Coordinator / Responsible Investigator Serap Ozmen and Associate Investigator Soner Sahin) will be blind; Researcher Ilknur Bostanci and assistant researcher Gulay Senel will appoint drugs and placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OM-85 (Active Comparator): OM-85 by mouth (3.5 mg once per day, first 10 days, consecutive 3 months; 10-10-10 days, standard treatment regimen) A second cure of treatment will be given 6 months after inclusion.
  Interventions: Biological: OM-85
- Placebo (Placebo Comparator): Placebo by mouth (Pregelatinized starch (Starch 1500)+Mannitol+Magnesium stearate+Anhydrous propyl gallate+Sodium glutamate) the same posology (3.5 mg once per day, first 10 days for consecutive 3 months) A second cure of treatment will be given 6 months after inclusion.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: OM-85 — OM-85 is an oral bacterial lysate of 21 different strains of 8 species and sub-species of the most common respiratory tract pathogens.
  Other Names: Vaxoral
  Arms: OM-85
Biological: Placebo — Pregelatinized starch (Starch 1500)+Mannitol+Magnesium stearate+Anhydrous propyl gallate+Sodium glutamate
  Arms: Placebo

SUMMARY:
Clinical research question: Can OM-85 reduce the recurrence of respiratory tract infections (RTIs) in children with AH by stimulating the immunological response of the host and therefore, as a consequence reduce the size of adenoid tissue in children with adenoid hypertrophy? Can this prevent further complications such as surgery need? Half of participants will receive OM-85, while other half will receive a placebo.

DETAILED DESCRIPTION:
OM-85 significantly reduces RTIs in children. This effect was proved by many clinical studies and meta-analyses. A Cochrane meta-analysis first published in 2006 and updated recently (Del-Rio-Navarro 2012) showed that immunostimulants (IS) could reduce acute RTIs (ARTIs) by almost 39% when compared to placebo. Among the different IS, OM-85 showed the most robust evidence with 4 trials of "A quality" according to the Cochrane grading criteria. Pooling six OM-85 studies, the Cochrane review reported a mean number of ARTIs reduction by -1.20 [95% Confidence Interval (CI): -1.75, -0.66 ] and a percentage difference in ARTIs by -35.9% [95% CI: -49.46, -22.35 ] compared to placebo.

Adenoid hypertrophy (AH) is one of the most important respiratory disease in preschool children. In normal conditions adenoid tissue enlarges up to 5 years and become smaller afterwards. But in some children who have recurrent upper respiratory tract infections (URTI)s, it keeps growing and this can be associated with complications. AH may cause recurrent respiratory infections and each infection contribute to enlargement of adenoid tissue thus promoting a vicious cycle. Additionally enlarged adenoids are known to be reservoir for microbes and cause of recurrent or long lasting RTIs.

AH is associated with chronic cough, recurrent and chronic sinusitis, recurrent tonsillitis, recurrent otitis media with effusion, recurrent other respiratory problems such as, nasal obstruction and sleep disturbances, sleep apneas. Eventually, AH causes loss of appetite and growth delay; it is often associated with misusing or over use of antibiotics and often eventually requires surgery. It decreases quality of life both in children and parents and it represents a burden not only for families but also for health care system and society due to increased health cost4.

In one study which investigated the structural and immunological aspects of tonsils and adenoids of 105 children (54 males and 51 females, aged between 4 and 18 years) who were affected by chronic inflammatory hypertrophy of palatine tonsils and adenoids which had not responded to previous medical treatments and who underwent adenotonsillectomy because of recurrent inflammatory episodes with fever, it was demonstrated that deficit in the activa-tion of the immune system could be represented by the small quan-tity of messenger ribonucleic acid (mRNA)s for interleukin-2 (IL-2) and interleukin-4 (IL-4) detected in our population, suggesting a defective activation of Th1 and Th2 lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* Children (age: 2-6 years)
* Who experienced recurrent RTIs (at least 3 episodes in 6 months before the inclusion)
* Who have symptoms of AH (snoring; mouth breathing awake; mouth breathing asleep; nasal congestion; hyponasal voice; chronic nasal discharge; daytime drowsiness, or hyperactivity; restless sleep; sleep apnoea <15 sec; night cough; and poor oral intake/weight loss) based on the symptoms score questionnaire

Exclusion Criteria:

* Atopy
* Gastroesophageal reflux
* Immune deficiency
* Asthma or allergic rhinitis
* Premature delivery
* Anatomic alterations of the respiratory tract; chronic respiratory diseases (tuberculosis and cystic fibrosis); autoimmune disease; liver
* Kidney failure; malnutrition; cancer
* Treatment with inhaled or systemic corticosteroids within the previous month
* Treatment with immunosuppressants, immunostimulants, gamma globulins, or anticonvulsive drugs within the previous 6 months.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of number of respiratory tract infections (RTIs) | within 12 months
  number of respiratory tract infections (RTIs) such as adenoiditis, sinusitis, tonsillitis, otitis, bronchitis

SECONDARY OUTCOMES:
Reduction in duration of RTIs | within 12 months
  duration of RTIs (day)
Reduction of antibiotic use | within 12 months
  number of antibiotic use
Reduction of missed school days | within 12 months
  missed school days (day)
Reduction of surgery need | within 12 months
  Whether or not surgery (adenoidectomy)
Adenoid and tonsil survey | within 12 months
  before and after the study
Size of adenoid tissue over the 12 months according to radiographic and flexible nasopharyngoscopic evaluation | 1 year
  The data will be recorded as a perceived percent obstruction of the choana by the adenoid pad, as seen through the endoscope; Lateral neck radiographs will taken and interpreted by the method of Cohen and Konak by a blinded radiologist (Cohen D, Konak S. The evaluation of radiographs of the nasopharynx. Clin Otolaryngol 1985; 10: 73-8.)

CONTACTS AND LOCATIONS:
Overall Officials: Serap Ozmen, Study Chair — Health of Science University, Dr Sami Ulus Maternity and Children Research and Training Hospital, Ankara, TURKEY

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (4):
  • Statistical Analysis Plan: SAP OM85adenoid (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT03243565/SAP_000.pdf
  • Informed Consent Form: ICF OM85adenoid (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT03243565/ICF_001.pdf
  • Study Protocol: SP OM85adenoid (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT03243565/Prot_002.pdf
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: SUM OM85adenoid (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT03243565/Prot_SAP_ICF_003.pdf